CLINICAL TRIAL: NCT05363657
Title: International REgistry of COnservative or Radical Treatment of Localized Kidney Tumors (i-RECORd)
Brief Title: International REgistry of COnservative or Radical Treatment of Localized Kidney Tumors
Acronym: i-RECORd
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: Società Italiana di Urologia (SIU) (Other); Italian Group for Advanced Laparo-Endoscopic and Robotic Urologic Surgery (AGILE) (Unknown)
Responsible Party: Principal Investigator, Andrea Minervini, Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: i-RECORd
Record Dates: First submitted 2022-03-14; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Partial Nephrectomy; Radical Nephrectomy; Ablation Techniques; Active Surveillance; Recurrence Free Survival; Watchful Waiting
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal tumor patiens: Patients with any renal tumor diagnosed with conventional imaging (computed tomography or magnetic resonance imaging) and undergoing to a clinical management in a hugh-volume center.
  Interventions: Procedure: Partial Nephrectomy (PN); Procedure: Radical Nephrectomy (RN); Procedure: Ablation therapy (AT); Diagnostic Test: Active Surveillance (AS)

INTERVENTIONS:
Procedure: Partial Nephrectomy (PN) — Conservative removal of kidney tumor. The procedure can be performed either with an open or laparoscopic or robotic approach.
Procedure: Radical Nephrectomy (RN) — Surgical removal of the affected kidney. Adrenal removal can be performed according to surgeon choice and clinical characteristics of the renal tumor. The procedure can be performed either with an open or laparoscopic or robotic approach.
Procedure: Ablation therapy (AT) — The procedure of tumor ablation performed with radiofrequency or cryoablation. The procedure can be performed either with a laparoscopic approach or percutaneous access.
Diagnostic Test: Active Surveillance (AS) — Active surveillance is defined as the initial management including the monitoring of renal tumor size by serial imaging with delayed treatment in case of progression.

SUMMARY:
Partial nephrectomy (PN) is the standard treatment for localized renal masses and should be preferred in clinical T1 (<7 cm tumor diameter) renal tumors over radical nephrectomy (RN) whenever technically feasible. Nonetheless, indications, approaches, techniques for PN, and correct reporting of outcomes, are still a matter of great debate within the urology community. Concurrently, case-report series suggested that alternative strategies for the treatment of localized renal tumors (ablation techniques (AT), watchful waiting (WW), active surveillance (AS)) could be feasible with acceptable oncologic outcomes in particular settings of patients with localized renal tumors. In this complex clinical scenario, the role surgeon-related and environmental factors (such as surgical experience, hospital resources, countries' social background and performance of health system) are important to address the best personalized approach in patients with renal tumors.

In the light of current evidence, many unsolved questions still remain and many unmet needs must be addressed. In particular, 1) the risk-benefit trade-offs between PN and RN for anatomically complex renal localized tumors; 2) the definition of evidence-based strategies to tailor the management strategy (AT vs WW vs AS vs surgery) in different subset of patients with particular clinical conditions (i.e. old, frail, comorbid patients); and 3) the definition of evidence-based recommendations to adapt surgical approach (open vs laparoscopic vs robotic) and resection techniques to different patient-, tumor-, and surgeon-specific characteristics.

To meet the challenges, to overcome the limitations of current kidney cancer literature (such as the retrospective study design, potential risk of biases, and heterogeneous follow-up of most series), and to provide high-quality evidence for future development of effective clinical practice Guidelines, we designed the international REgistry of COnservative or Radical treatment of localized kiDney tumors (i-RECORD) Project.

The expected impact of the i-RECORD project is to provide robust evidence on the leading clinical and environmental factors driving selection of the management strategy in patients with kidney cancer, and the differential impact of different management strategies (including AS, WW, AT, PN and RN) on functional, perioperative and oncological outcomes, as well as quality of life assessment, at a mid-long term follow-up (5-10 years).

DETAILED DESCRIPTION:
Study design

The overall objective of the i-RECORD project is to build a multicentre multi-arm multi-stage prospective observational registry collecting data on the management of kidney cancer in consecutive patients treated at 50 tertiary referral Centers worldwide over a 2 years-period and with 5 years of follow-up

. On this registry, six prospective trials with specific objectives have been built.

The i-RECORd project is designed as an observational prospective longitudinal trial involving 50 international, very-high-volume tertiary referral Centers with extensive experience in management of kidney cancer. Centers will be included in the project only if they will be able to certify at least to: 1) perform 150 partial and radical nephrectomy/year, or 2) to perform 80 ATs/year, or 3) to include 50 patients in WW/AS protocols/year.

The enrollment and follow-up periods will be 2 and 5 years, respectively. The estimate of patients' enrollment over the study period is 10'000 inclusions.

The 50 Centers finally enrolled in the i-RECORD project will be given the access to a web-based platform for data collection for 24 months from the starting date of the project.

A web-based e-form platform will be used for data collection.

Data collection

This observational study aims to obtain controlled, qualitative and quantitative, data of the enrolled patients through a web-based e-form platform. For all patients it will be asked to complete a data collection form specifically designed for this study, consisting of some subfolders:

1. Anthropometric, pre-operative and comorbidity data (patient characteristics).
2. Imaging data e and pre-operative tumor features (tumor characteristics).
3. Intra-operative and post-operative data (treatment characteristics).
4. Histopathological analysis (tumor histopathological characteristics).
5. Patients follow-up variables (at 6, 12, 24 and 60 months from the treatment) (follow-up characteristics).

Decision Analysis Modeling

Beyond traditional descriptive and inferential statistical analyses, the i-RECORd project will provide a comprehensive overview of the current selection criteria for each type of management option by applying innovative statistical methods (Decision Analysis Modeling through discrete choice models) to determine the differential impact of all potential relevant variables on the choice of treatment. To do so, we will consider specific clinical scenarios (clinical clusters) made of the integration of patient characteristics (comorbidity score, performance status, age, gender, etc.), patient-reported outcomes measures (PROMs), tumors anatomical features (degree of complexity, clinical diameter, side, location within the kidney, involvement of renal sinus or collecting system, etc.), surgeon-related factors (surgical experience and background), hospital economic availabilities (i.e. open, laparoscopic, robotic surgery) and other country-specific socio-economical features in order to determine the impact of such variables on the final choice of treatment.

By applying the discrete choice model to the analysis of the prospective dataset, the i-RECORd project will overcome the current state of the art in the treatment of localized renal tumors as it will show how the choice of treatment is performed by the decision-maker (at a surgeon- and hospital-level) in each specific clinical cluster of patients, why that choice was performed according to a careful analysis of the personalized patient setting and whether that choice will influence the postoperative outcomes.

Adapted MAMS Registry

The i-RECORD will be designed adapting the innovative concept of multi-arm, multi-stage (MAMS) platform randomized trials (used, for instance, for the design of the Systemic Therapy in Advancing or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) Trial) to create a dynamic, observational registry evaluating simultaneously different management options in different patient- and/or tumor-related scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of renal tumor susceptible to active treatment or AS/WW.
* Age ≥18 years
* Informed consent signed

Exclusion Criteria:

* Patient refuse to participate in clinical research.
* Urothelial renal carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population include patients with a radiological diagnosis of kidney tumor susceptible to surgical treatment (RN or PN) or AT or WW/AS will be eligible.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To test the effectiveness of partial nephrectomy for the treatment of localized renal tumors (T1-T2N0M0) with regards to recurrence-free survival and cardiovascular accidents and mortality in comparison to radical nephrectomy? | Assesments of the outcome at 60 months from the surgical intervention. Time frame : 5 years
  The preoperative characteristics of the patients will be specifically evaluated to calculate any heterogeneity between the two groups. In detail, anthropometric and comorbidity features, previous abdominal surgery, blood chemistry values, blood pressure, smoking habit, preoperative life expectancy, and frailty grade will be assessed. Imaging features of the tumor will be considered, including the characteristics necessary for the calculation of the PADUA, R.E.N.A.L., and Contact-Surface-Area scores. Patients with a node-positive or metastatic disease diagnosed with conventional imaging (CT scan/MRI) will be excluded. Intra-operative and post-operative outcomes will be evaluated. Histopathological features of the tumor will be assessed.
  Patients will be followed up with conventional imaging according to the International guidelines (ultrasound, CT, MRI). Serum creatinine, platelets and estimated glomerular function (eGFR), the onset of cardiovascular adverse events will be registered.
To test the effectiveness of robotic approach in partial nephrectomy to increase the "Trifecta" rate after nephron-sparing surgery in patients with T1-T2N0M0 renal tumors. | Assesment of the "Trifecta" outcome will be performed at 12 months from the surgical intervention. Time frame: 1 year.
  "Trifecta" rate is defined as 1) Absence of intraoperative and postoperative surgical complications; 2) absence of positive surgical margins or recurrences on tumor resection site during a 5-year follow-up; 3) Absence of clinically significant renal function loss at one year after surgery. Renal function will be evaluated using the estimated glomerular filtration rate (eGFR) in ml/min/1.73 m^2 using the CKD-EPI Creatinine Equation (2021). A clinically significant loss will be considered if >25% from eGFR at baseline.
  The "Trifecta" outcome will be evaluated one year from surgery.

SECONDARY OUTCOMES:
To evaluate the differential impact of patients' comorbidities, tumors' complexity, surgeons' experience, country-related socio-cultural factors and hospital financial resources on the selection of the type of clinical management. | Assesment will be done at the time of registering the type of surgery/clinical managing adopted. Time frame: <1 week from patients accrual..
  The following variables will be evaluated:
  1. Anthropometric, pre-operative and comorbidity data (patient characteristics).
  2. Imaging data and pre-operative tumor features (tumor characteristics).
  3. Centre facilities (laparoscopic/robot assisted, interventional radiology) , volume centre (PN/RN ratio, availability of Multidisciplinary Tumor Board)
  4. Intra-operative and post-operative data (treatment characteristics).
  5. Histopathological analysis (tumor histopathological characteristics). The outcome will be considered as the type of clinical management selected: active surveillance (AS) vs ablative treatment (AT) vs partial nephrectomy (PN) vs radical nephrectomy (RN).
To evaluate the impact of the antiaggregant and/or antiplatelet treatment at baseline and during partial nephrectomy on hemorrhagic complications. | Outcome assesment will be done at 90 days from surgery. Time frame: 3 months
  The eventual anticoagulant therapy (heparin, warfarin, enoxaparin, fondaparinux) and/or antiplatelet therapy (clopidogrel, ticagrelor, prasugrel, dipyridamole, dipyridamole/aspirin, ticlopidine, eptifibatide) use in patients at baseline and at time of surgery will be assessed.
  Hemorrhagic complications (graded according to the "Clavien-Dindo classification") will be evaluated during surgery (intraoperative) and within 90 days (postoperative) with particular attention to the management of hemorrhage (patient monitoring, transfusion, selective embolization, re-intervention with/without kidney removal).
To assess in patients with antiaggregant and/or antiplatelet treatment at baseline any potential change of this therapy at the time of treatment associated with the absence of hemorrhagic complications. | Outcome assesment will be done at 90 days from surgery. Time frame: 3 months
  The eventual anticoagulant therapy (heparin, warfarin, NAO, enoxaparin, fondaparinux) and/or antiplatelet therapy (clopidogrel, ticagrelor, prasugrel, dipyridamole, dipyridamole/aspirin, ticlopidine, eptifibatide) use in patients at baseline and at time of surgery will be assessed.
  Change of treatment from baseline to time of surgery will be considered and specifically evaluated according to the underlying cardio- and/or peripheral- and/or cerebro-vascular diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Minervini, Prof., Principal Investigator — Dipartimento di Medicina Clinica e Sperimentale Via o Piazza Largo Brambilla 3 - 50134 Firenze (Italy)
Locations (37):
- United States (7):
  - Institute of Urology, University of Southern California., Los Angeles, California
  - University of California San Diego, Moores Cancer Center, San Diego, California
  - Stanford University, Stanford, California
  - Loyola University Medical Center, Edward Hines VA Hospital, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - VCU Health System, Richmond, Virginia
  - Swedish Hospital, Seattle, Washington
- Medical University of Vienna, Vienna General Hospital, Vienna, Austria
- Belgium (3):
  - University of Bruxelles, Brussels
  - University Hospitals Leuven, Leuven
  - Onze Lieve Vrouw Hospital, Leuven
- Santa Casa da Misericórdia de Fortaleza, Fortaleza, Brazil
- University of Patras, Pátrai, Greece
- Italy (14):
  - Urology, Andrology & Kidney Transplantation Unit, University of Bari, Bari
  - Policlinico S. Orsola Malpighi, Bologna
  - Department of Urology, University of Florence, Unit of Oncologic Minimally-Invasive Urology and Andrology, Careggi Hospital, Florence
  - Policlinico Riuniti, Università di Foggia., Foggia
  - Division of Urology, University of Genoa,Policlinico San Martino Hospital, Genova
  - Azienda Ospedaliera Policlinico "G. Martino", Università di Messina., Messina
  - San Raffaele Scientific Institute, Milan, Italy; Division of Experimental Oncology/Unit of Urology, URI, IRCCS San Raffaele Hospital, Milan
  - Policlinico Istituto Europeo di Oncologia (IEO), Milan
  - Istituto Nazionale dei Tumori Fondazione Senatore "G. Pascale", Napoli
  - Institute Oncology Veneto (IOV), Padua
  - Humanitas Hospital, Rozzano
  - Università degli Studi di Torino, Ospedale S. Luigi Gonzaga., Torino
  - Università degli studi di Torino, Ospedale Molinette, Torino
  - AOUI Verona, Verona
- Jikei University School of Medicine, Tokyo, Japan
- Amsterdam University Medical Centers, Amsterdam, Netherlands
- Poland (2):
  - European Health Center, Otwock
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Warsaw
- N.N. Blokhin National Medical Research Center of Oncology, Moscow, Russia
- NG Teng Fong General Hospital, Singapore, Singapore
- Spain (2):
  - Fundaciò Puigvert, Barcelona
  - Hospital Universitario Ramón y Cajal, University of Alcalá, Madrid
- United Kingdom (2):
  - Bristol Urological Institute, Bristol
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The study protocol has been shared on the web platform of the i-RECORd project. The study has been shared with a specific Twitter page for the study.
Supporting Information: Study Protocol
Time Frame: The data will be available after Clinical.trial.gov study acceptance
Access Criteria: Access to the study protocol will be free to any researcher.
URL: https://twitter.com/iRECORdProject

REFERENCES:
- [Result] Ljungberg B, Bensalah K, Canfield S, Dabestani S, Hofmann F, Hora M, Kuczyk MA, Lam T, Marconi L, Merseburger AS, Mulders P, Powles T, Staehler M, Volpe A, Bex A. EAU guidelines on renal cell carcinoma: 2014 update. Eur Urol. 2015 May;67(5):913-24. doi: 10.1016/j.eururo.2015.01.005. Epub 2015 Jan 21. PMID 25616710
- [Result] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Allen C, Barber RM, Barregard L, Bhutta ZA, Brenner H, Dicker DJ, Chimed-Orchir O, Dandona R, Dandona L, Fleming T, Forouzanfar MH, Hancock J, Hay RJ, Hunter-Merrill R, Huynh C, Hosgood HD, Johnson CO, Jonas JB, Khubchandani J, Kumar GA, Kutz M, Lan Q, Larson HJ, Liang X, Lim SS, Lopez AD, MacIntyre MF, Marczak L, Marquez N, Mokdad AH, Pinho C, Pourmalek F, Salomon JA, Sanabria JR, Sandar L, Sartorius B, Schwartz SM, Shackelford KA, Shibuya K, Stanaway J, Steiner C, Sun J, Takahashi K, Vollset SE, Vos T, Wagner JA, Wang H, Westerman R, Zeeb H, Zoeckler L, Abd-Allah F, Ahmed MB, Alabed S, Alam NK, Aldhahri SF, Alem G, Alemayohu MA, Ali R, Al-Raddadi R, Amare A, Amoako Y, Artaman A, Asayesh H, Atnafu N, Awasthi A, Saleem HB, Barac A, Bedi N, Bensenor I, Berhane A, Bernabe E, Betsu B, Binagwaho A, Boneya D, Campos-Nonato I, Castaneda-Orjuela C, Catala-Lopez F, Chiang P, Chibueze C, Chitheer A, Choi JY, Cowie B, Damtew S, das Neves J, Dey S, Dharmaratne S, Dhillon P, Ding E, Driscoll T, Ekwueme D, Endries AY, Farvid M, Farzadfar F, Fernandes J, Fischer F, G/Hiwot TT, Gebru A, Gopalani S, Hailu A, Horino M, Horita N, Husseini A, Huybrechts I, Inoue M, Islami F, Jakovljevic M, James S, Javanbakht M, Jee SH, Kasaeian A, Kedir MS, Khader YS, Khang YH, Kim D, Leigh J, Linn S, Lunevicius R, El Razek HMA, Malekzadeh R, Malta DC, Marcenes W, Markos D, Melaku YA, Meles KG, Mendoza W, Mengiste DT, Meretoja TJ, Miller TR, Mohammad KA, Mohammadi A, Mohammed S, Moradi-Lakeh M, Nagel G, Nand D, Le Nguyen Q, Nolte S, Ogbo FA, Oladimeji KE, Oren E, Pa M, Park EK, Pereira DM, Plass D, Qorbani M, Radfar A, Rafay A, Rahman M, Rana SM, Soreide K, Satpathy M, Sawhney M, Sepanlou SG, Shaikh MA, She J, Shiue I, Shore HR, Shrime MG, So S, Soneji S, Stathopoulou V, Stroumpoulis K, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tadese F, Tedla BA, Tessema GA, Thakur JS, Tran BX, Ukwaja KN, Uzochukwu BSC, Vlassov VV, Weiderpass E, Wubshet Terefe M, Yebyo HG, Yimam HH, Yonemoto N, Younis MZ, Yu C, Zaidi Z, Zaki MES, Zenebe ZM, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-years for 32 Cancer Groups, 1990 to 2015: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2017 Apr 1;3(4):524-548. doi: 10.1001/jamaoncol.2016.5688. PMID 27918777
- [Result] Campbell S, Uzzo RG, Allaf ME, Bass EB, Cadeddu JA, Chang A, Clark PE, Davis BJ, Derweesh IH, Giambarresi L, Gervais DA, Hu SL, Lane BR, Leibovich BC, Pierorazio PM. Renal Mass and Localized Renal Cancer: AUA Guideline. J Urol. 2017 Sep;198(3):520-529. doi: 10.1016/j.juro.2017.04.100. Epub 2017 May 4. PMID 28479239
- [Result] Stewart SB, Thompson RH, Psutka SP, Cheville JC, Lohse CM, Boorjian SA, Leibovich BC. Evaluation of the National Comprehensive Cancer Network and American Urological Association renal cell carcinoma surveillance guidelines. J Clin Oncol. 2014 Dec 20;32(36):4059-65. doi: 10.1200/JCO.2014.56.5416. Epub 2014 Nov 17. PMID 25403213
- [Result] Motzer RJ, Jonasch E, Agarwal N, Bhayani S, Bro WP, Chang SS, Choueiri TK, Costello BA, Derweesh IH, Fishman M, Gallagher TH, Gore JL, Hancock SL, Harrison MR, Kim W, Kyriakopoulos C, LaGrange C, Lam ET, Lau C, Michaelson MD, Olencki T, Pierorazio PM, Plimack ER, Redman BG, Shuch B, Somer B, Sonpavde G, Sosman J, Dwyer M, Kumar R. Kidney Cancer, Version 2.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Jun;15(6):804-834. doi: 10.6004/jnccn.2017.0100. PMID 28596261
- [Result] Volpe A, Blute ML, Ficarra V, Gill IS, Kutikov A, Porpiglia F, Rogers C, Touijer KA, Van Poppel H, Thompson RH. Renal Ischemia and Function After Partial Nephrectomy: A Collaborative Review of the Literature. Eur Urol. 2015 Jul;68(1):61-74. doi: 10.1016/j.eururo.2015.01.025. Epub 2015 Feb 20. PMID 25703575
- [Result] Finelli A, Ismaila N, Bro B, Durack J, Eggener S, Evans A, Gill I, Graham D, Huang W, Jewett MA, Latcha S, Lowrance W, Rosner M, Shayegan B, Thompson RH, Uzzo R, Russo P. Management of Small Renal Masses: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2017 Feb 20;35(6):668-680. doi: 10.1200/JCO.2016.69.9645. Epub 2017 Jan 17. PMID 28095147
- [Result] Larcher A, Sun M, Dell'Oglio P, Trudeau V, Boehm K, Schiffmann J, Tian Z, Fossati N, Capitanio U, Briganti A, Montorsi F, Karakiewicz P. Mortality, morbidity and healthcare expenditures after local tumour ablation or partial nephrectomy for T1A kidney cancer. Eur J Surg Oncol. 2017 Apr;43(4):815-822. doi: 10.1016/j.ejso.2016.08.023. Epub 2016 Sep 17. PMID 27692535
- [Result] Larcher A, Fossati N, Tian Z, Boehm K, Meskawi M, Valdivieso R, Trudeau V, Dell'Oglio P, Buffi N, Montorsi F, Guazzoni G, Sun M, Karakiewicz PI. Prediction of Complications Following Partial Nephrectomy: Implications for Ablative Techniques Candidates. Eur Urol. 2016 Apr;69(4):676-682. doi: 10.1016/j.eururo.2015.07.003. Epub 2015 Jul 21. PMID 26206408
- [Result] Kim SP, Campbell SC, Gill I, Lane BR, Van Poppel H, Smaldone MC, Volpe A, Kutikov A. Collaborative Review of Risk Benefit Trade-offs Between Partial and Radical Nephrectomy in the Management of Anatomically Complex Renal Masses. Eur Urol. 2017 Jul;72(1):64-75. doi: 10.1016/j.eururo.2016.11.038. Epub 2016 Dec 14. PMID 27988238
- [Result] Patel HD, Pierorazio PM, Johnson MH, Sharma R, Iyoha E, Allaf ME, Bass EB, Sozio SM. Renal Functional Outcomes after Surgery, Ablation, and Active Surveillance of Localized Renal Tumors: A Systematic Review and Meta-Analysis. Clin J Am Soc Nephrol. 2017 Jul 7;12(7):1057-1069. doi: 10.2215/CJN.11941116. Epub 2017 May 8. PMID 28483780
- [Result] Mari A, Campi R, Schiavina R, Amparore D, Antonelli A, Artibani W, Barale M, Bertini R, Borghesi M, Bove P, Brunocilla E, Capitanio U, Da Pozzo L, Daja J, Gontero P, Larcher A, Li Marzi V, Longo N, Mirone V, Montanari E, Pisano F, Porpiglia F, Simeone C, Siracusano S, Tellini R, Trombetta C, Volpe A, Ficarra V, Carini M, Minervini A; Collaborators. Nomogram for predicting the likelihood of postoperative surgical complications in patients treated with partial nephrectomy: a prospective multicentre observational study (the RECORd 2 project). BJU Int. 2019 Jul;124(1):93-102. doi: 10.1111/bju.14680. Epub 2019 Feb 12. PMID 30653796
- [Result] Psutka SP, Leibovich BC. Management of inferior vena cava tumor thrombus in locally advanced renal cell carcinoma. Ther Adv Urol. 2015 Aug;7(4):216-29. doi: 10.1177/1756287215576443. PMID 26445601
- [Result] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Result] Sydes MR, Parmar MK, Mason MD, Clarke NW, Amos C, Anderson J, de Bono J, Dearnaley DP, Dwyer J, Green C, Jovic G, Ritchie AW, Russell JM, Sanders K, Thalmann G, James ND. Flexible trial design in practice - stopping arms for lack-of-benefit and adding research arms mid-trial in STAMPEDE: a multi-arm multi-stage randomized controlled trial. Trials. 2012 Sep 15;13:168. doi: 10.1186/1745-6215-13-168. PMID 22978443